CLINICAL TRIAL: NCT06870734
Title: General Anesthesia Versus Loco-Regional Anesthesia for Transcarotid Trancatheter Aortic Valve Replacement - a Retrospective Cohort Study
Brief Title: General Anesthesia Versus Loco-Regional Anesthesia for Transcarotid Trancatheter Aortic Valve Replacement
Acronym: GALATTAVI
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Richard DESCAMPS, Doctor, University Hospital, Caen
Other Study IDs: 2024102821344400000170001538
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Aortic Stenosis
Keywords: general anesthesia; cervical block; locoregional anesthesia; TAVR; cardiovascvular intervention
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- General anesthesia: Patients undergoing transcarotid transaortic valve replacement under general anesthesia
- Regional anesthesia: Patients undergoing transcarotid transaortic valve replacement under regional anesthesia

SUMMARY:
Transcarotid transcatheter aortic valve replacement (Transcarotid TAVR) has been increasingly used as an alternative to the transfemoral approach. The general anesthesia, locoragional anesthesia or local anesthesia are three anesthesia techniques that can be used for transcarotid TAVR. We aim to compare the locoregional approach to gerneral anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent a transcarotid TAVR at the University Hospital of Caen between October 2021 (when the first TAVR was performed under locoregional anesthesia) and December 2024

Exclusion Criteria:

* Patient's refusal to allow data collection and lack of data regarding the primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent a transcarotid TAVR at the University Hospital of Caen between October 2021 (when the first TAVR was performed under locoregional anesthesia) and December 2024
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2025-03-07 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | 7 days
  Composite endpoint combining mortality and stroke in the first post-operative week

SECONDARY OUTCOMES:
Death | 7 days
  Death occuring during the first week after intervention
Stroke | 7 days
  Stroke occuring during the first week after the intervention
30 day mortality | 30 days
  Death occuring during the first month after intervention
1 year mortality | 1 year
  Death occuring during the first year after intervention
Vasopressive drugs | 1 day
  Use of vasopressive drugs during the intervention

OTHER OUTCOMES:
Pacemaker implantation | 7 to 30 days
  Pacemaker implantation during the index hospitalisation

IPD SHARING:
Plan to Share IPD: Undecided